CLINICAL TRIAL: NCT05126732
Title: Is Ganglion Cell Thickness the Main Problem in Enuresis Nocturna?
Brief Title: Ganglion Cell Thickness in Enuresis Nocturna
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Yasar Issi, Asistant Professor, Izmir Bakircay University
Other Study IDs: 341/321
Record Dates: First submitted 2021-10-28; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Enuresis, Nocturnal; Ganglion; Circadian Rhythm Disorders
Keywords: enuresis; optical coherence tomography
MeSH Terms: conditions — Nocturnal Enuresis; Ganglion Cysts; Chronobiology Disorders; Enuresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The precise role of the intrinsic circadian regulatory mechanism behind the pathogenesis of enuresis is not fully understood, but in theory, circadian rhythm irregularity may be the primary pathogenic mechanism not only for urinary outflow mechanisms but also for nocturnal bladder function. The proximity between SCN centers that control AVP release, sleep/arousal, voiding, and baroreregulation may provide the basis for circadian rhythm disturbance in one or more of these biological functions. Ganglion cells containing melanopsin pigment in the retina transmit the information they receive from the outside world about the light-dark state to the SCN via the retinohypothalamic pathway. Peripapillary retinal nerve fiber layer (RNFL) thickness, optic nerve head and macula are examined most frequently for the diagnosis of glaucoma and the detection of progression with optical coherence tomography (OCT). If differences in ganglion cell thickness can be detected using OCT in these children, a new avenue in Enuresis Nocturna may be opened.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 5-18
* have enuresis

Exclusion Criteria:

* have any eye conditions

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients aged 5-18 years, with enuresis, without any eye disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Difference in ganglion cell thickness in enuretic children | Baseline
  Normal values in RNFL measurements on OCT 75 (lowest)-107.2 (highest)

CONTACTS AND LOCATIONS:
Locations (1):
- Bakircay University, Izmir, Turkey (Türkiye)